CLINICAL TRIAL: NCT00796692
Title: Efficacy and Safety of Body Weight Adjusted Nadroparin vs Standard Unfractionated Heparin for the Initial Treatment of Pulmonary Thromboembolism：a Multi-Centre, Randomised Controlled Trial in China
Brief Title: Nadroparin for the Initial Treatment of Pulmonary Thromboembolism
Acronym: NATSPUTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Professor Chen WANG, Beijing Institute of Respiratory Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA703B07; 2001BA703B13
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Pulmonary Embolism; Thromboembolism; Vascular Diseases; Thrombosis
Keywords: Heparin; Low molecular weight heparin; Safety; Efficacy; Cost effective
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism; Vascular Diseases; Thrombosis | interventions — Nadroparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): Low molecular weight heparin
  Interventions: Drug: Nadroparin
- Group 1 (Active Comparator): Unfractionated heparin(UFH)
  Interventions: Drug: Unfractionated heparin(UFH)

INTERVENTIONS:
Drug: Nadroparin — LMWH is given with a weight adjusted dose of 86 international anti-factor Xa units of nadroparin (Fraxiparine) per kilogram of body weight(86 anti-factor Xa IU/kg) subcutaneously every 12 hours,which will be used at least 5-7 days.
  Other Names: Low moleculor weight hepatin
  Arms: Group 2
Drug: Unfractionated heparin(UFH) — UFH is received with an initial bolus dose of 80 IU per kilogram, followed by a continuous intravenous infusion at an initial rate of 18 IU per kilogram per hour. The dose is subsequently adjusted so that the activated partial thromboplastin time (APTT) would be 1.5 to 2.5 times the control value in normal subjects. The tests are performed 4 hours after the start of treatment, whenever a sub-therapeutic APTT had been measured after a dose adjustment, and otherwise daily.UFH will be used at least 5-7 days.
  Other Names: Standard Unfractionated heparin
  Arms: Group 1

SUMMARY:
Low-molecular-weight heparin (LWMH) appears to be at least as effective and safe as standard, unfractionated heparin (UFH)for the treatment of patients with deep vein thrombosis(DVT) and may also be so in patients with pulmonary thromboembolism (PTE). Only limited data are available on the evaluation of body weight adjusted LWMH and standard UFH for the initial treatment of PTE in Chinese population. The aim of this study is to determine whether body weight-adjusted, subcutaneous Nadroparin is as effective and safe as UFH for treatment of patients with objectively documented PTE.

DETAILED DESCRIPTION:
Low-molecular-weight heparin (LWMH) appears to be at least as effective and safe as standard, unfractionated heparin (UFH)for the treatment of patients with deep vein thrombosis(DVT) and may also be so in patients with pulmonary thromboembolism (PTE). Only limited data are available on the evaluation of body weight adjusted LWMH and standard UFH for the initial treatment of PTE in Chinese population.

The aim of this study is to determine whether body weight-adjusted, subcutaneous Nadroparin is as effective and safe as UFH for treatment of patients with objectively documented PTE.

An open-label, adjudicator-blinded, randomized controlled trial of patients with symptomatic non-massive PTE from 37 major hospitals in China is conducted . Intravenous UFH was administered received an initial bolus dose of 80 IU/kg, followed by a continuous infusion at an initial rate of 18 IU/kg /hour. The dose was subsequently adjusted by activated partial thromboplastin time (APTT) monitoring. LMWH (nadroparin) was administered subcutaneously at a dose of 86 anti-factor Xa IU/kg every 12 hours.

Both treatments were overlapped with at least 3 months of warfarin therapy. Main outcome measures were combined end point of clinical effect, image improvement,Recurrent venous thromboembolism(VTE), major bleeding, and death within 14 days and 3 months of randomization.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Symptomatic non massive PTE confirmed either by a high probability ventilation-perfusion lung scanning (V/Q scan) or by the presence of intraluminal filling defect on spiral computed tomographic pulmonary angiography (CTPA)
* Haemodynamic stabile, anatomic obstruction no more than 2 lobes on CTPA, or defect no more than 7 segments on V/Q scan,and normal right ventricular function
* Symptoms within 15 days
* Written informed consent obtained before randomization.

Exclusion Criteria:

* Unfractioned heparin anticoagulation for more than 36 hours prior enrollment,
* Massive PTE or sub-massive PTE requiring thrombolytic therapy or pulmonary embolectomy; Active bleeding or disorders contraindicating anticoagulant therapy
* Chronic thromboembolism pulmonary hypertension(CTEPH) without evidence of recent episode; Severe hepatic or renal failure
* Allergy to heparin, other components of Tinzaparin or acenocoumarol,
* Pregnant status;a life expectancy of less than 3 months;
* Previous thrombocytopenia induced by heparin
* Thrombocytopenia < 100000/mm3,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2002-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Clinical and image(including V/Q scan and CTPA) improvement | Time Frame: 14days

SECONDARY OUTCOMES:
Recurrent venous thromboembolism(VTE), major bleeding death Heparin-induced thrombocytopenia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen WANG, Prof, Principal Investigator — Beijing Institute of Respiratory Medicine,Beijing Chao Yang Hospital
Locations (39):
- China (39):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing General Hospital of the Air-force PLA, Beijing, Beijing Municipality
  - Beijing Naval General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing No 6 Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou, Guandong
  - Guangzhou Institute of Respiratory Disease，Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Worker's Hospital, Hebei Medical University, Tangshan, Hebei
  - The Affiliated Hospital of Hubei Coal University, Tangshan, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Liaoning Angang Tiedong Hospital, Anshan, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The General Hospital of Shenyang Military Command, Shenyang, Liaoning
  - The Affiliated Hospital of Shenyang Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Medical College Jining, Jining, Shandong
  - The Affiliated Hospital of Medical College Qingdao, Qingdao, Shandong
  - Shandong Yantaishan Hospital, Yantai, Shandong
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital(8), Shanghai, Shanghai Municipality
  - Shanxi Datong 5th Hospital, Datong, Shanxi
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Thoracic Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Xinjiang People's Hospital, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Affiliated with Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Background] Pang BS, Wang C, Lu Y, Yang YH, Xing GH, Mao YL, Huang XX, Zhai ZG. [Changes of blood coagulative and fibrinolytic system and function of pulmonary vascular endothelium after therapy in patients with acute pulmonary thromboembolism]. Zhonghua Yi Xue Za Zhi. 2007 Nov 20;87(43):3074-8. Chinese. PMID 18261355
- [Background] Zhu L, Yang Y, Wu Y, Zhai Z, Wang C. Value of right ventricular dysfunction for prognosis in pulmonary embolism. Int J Cardiol. 2008 Jun 23;127(1):40-5. doi: 10.1016/j.ijcard.2007.06.093. Epub 2007 Aug 22. PMID 17716753
- [Background] Zhu L, Wang C, Yang Y, Wu Y, Zhai Z, Dai H, Pang B, Tong Z. Value of transthoracic echocardiography in therapy regimens evaluation in pulmonary embolism. J Thromb Thrombolysis. 2008 Dec;26(3):251-6. doi: 10.1007/s11239-007-0087-8. Epub 2007 Aug 21. PMID 17705052
- [Background] Liu CP, Lu WX, Liu WG, Chen HW, Wang C. [The low molecular weight heparin on rat pulmonary surfactant associated protein A of acute pulmonary embolism]. Zhonghua Yi Xue Za Zhi. 2007 Mar 6;87(9):634-6. Chinese. PMID 17550736
- [Background] Zhu L, Yang YH, Wu YF, Zhai ZG, Wang C; National Project of the Diagnosis and Treatment Strategies for Pulmonary Thromboembolism investigators. Value of transthoracic echocardiography combined with cardiac troponin I in risk stratification in acute pulmonary thromboembolism. Chin Med J (Engl). 2007 Jan 5;120(1):17-21. PMID 17254482
- [Background] Sun KK, Wang C, Guli XT, Luo Q. [Risk factors and clinical features of deep venous thrombosis: a report of 388 cases]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Nov;27(11):727-30. Chinese. PMID 15634380
- [Background] Zhai ZG, Wang C, Liu YM, Qin ZQ. [Comparison of unfractionated heparin and low molecular weight heparin in pulmonary thromboembolism: meta-analysis]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2004 Jun;26(3):221-6. Chinese. PMID 15266820
- [Background] Pang BS, Wang C, Luo Q, Zhang LM, Zhu M, Mao YL, Huang XX, Guo WJ. [Study of the function of coagulation, fibrinolysis and pulmonary vascular endothelium before and after experimental pulmonary thromboembolism in rabbits]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Jun;27(6):381-4. Chinese. PMID 15256085
- [Background] Zai ZG, Wang C. [Advances in the study of pulmonary thromboembolism]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Jan;27(1):14-8. No abstract available. Chinese. PMID 14989818
- [Background] Qin ZQ, Wang C. [Comparison of thrombolysis and anticoagulation in pulmonary thromboembolism: a meta-analysis]. Zhonghua Jie He He Hu Xi Za Zhi. 2003 Dec;26(12):772-5. Chinese. PMID 14720434